CLINICAL TRIAL: NCT06088875
Title: Nebulization Versus Spray-as-You-Go Airway Topical Anesthesia Using Dexmedetomidine and Lidocaine Mixture During Awake Flexible Fiberoptic Intubation in Temporomandibular Ankylosis: A Randomized Double-Blind Trial
Brief Title: Nebulization Versus Spray-as-You-Go Airway Topical Anesthesia Using Dexmedetomidine and Lidocaine Mixture During Awake Flexible Fiberoptic Intubation in Temporomandibular Ankylosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mahmoud Hassan El-Baradei, Resident of Anesthesiology, Surgical Intensive Care and Pain Medicine, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 36264MS159/4/23
Record Dates: First submitted 2023-10-03; First posted 2023-10-18 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Nebulization; Spray-as-You-Go; Dexmedetomidine; Lidocaine; Temporomandibular Ankylosis
MeSH Terms: conditions — Temporomandibular ankylosis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group N (Nebulization group) (Experimental): Patients will receive a mixture of 2% lidocaine 10 ml and dexmedetomidine 1 μg/kg nebulization + saline 10 ml via spray-as-you-go technique.
  Interventions: Drug: Nebulization
- Group S (Spray-as-you-go) (Experimental): Patients will receive a mixture of 2% lidocaine 10 ml and dexmedetomidine 1 μg/kg via spray-as-you-go technique + saline 10 ml nebulization.
  Interventions: Drug: Spray-as-you-go

INTERVENTIONS:
Drug: Nebulization — Patients will be nebulized with mixture of 2% lidocaine 10 ml and dexmedetomidine 1 μg/kg by using wall nebulizer for 15 min before awake fiberoptic intubation. Patients in group S will receive saline 10 ml nebulization
  Arms: Group N (Nebulization group)
Drug: Spray-as-you-go — Patients will receive a mixture of 2% lidocaine 10 ml and dexmedetomidine 1 μg/kg via spray-as-you-go technique + saline 10 ml nebulization. Patients in group N will receive saline via spray-as-you-go technique
  Arms: Group S (Spray-as-you-go)

SUMMARY:
The aim of this study is to compare the efficacy of airway topical anesthesia with nebulization to the spray-as-you-go technique using dexmedetomidine and lidocaine mixture to achieve upper airway anesthesia in TMJ ankylosis patients.

DETAILED DESCRIPTION:
Awake fiber-optic intubation (AFOI) has become the accepted gold standard technique for management of recognized difficult airway as the larynx remains in a posterior position and the patient is able to protect the airway from soiling and can maintain the airway patency as well as spontaneous breathing efforts. Awake intubation requires that the patient remains calm and cooperative and is provided with sufficient anxiolysis, analgesia, and topical anesthesia without compromising the airway.

Gag reflex, cough, and laryngospasm can be upsetting during the process. Awake patients never permit airway instrumentation without airway anesthesia. Therefore, effective airway anesthesia is required for airway instrumentation and patient comfort.

For awake intubation, topical airway anesthesia can be provided either by using fiberoptic bronchoscope (FOB) to apply local anaesethic to the airway by a "spray-as-you-go" technique or nebulizing the patient for about 10-15 min.

ELIGIBILITY:
Inclusion Criteria:

* Age from 21to 65 years.
* Both sexes.
* American Society of Anesthesiologists (ASA) physical status I or II and scheduled for elective surgery requiring general anesthesia , and known to have Temporomandibular joint ankylosis and expected to be difficult intubation patient due to restriction of jaw mobility and limited mouth opening less than 2 fingers.

Exclusion Criteria:

* History of allergy to dexmedetomidine or lidocaine.
* History of drug abuse.
* Concomitant use of medications which may exaggerate the heart rate (HR) response of -dexmedetomidine (e.g. digoxin or β-adrenergic antagonists), HR <50 beats/min, systolic blood pressure (SBP) <90 mmHg.
* Pregnancy.
* Morbid obesity( BMI more than 35).
* Patients on anticoagulants, nasal trauma, deformity or polyp, CSF rhinorrhea, fracture base skull.
* Cardiac and/or respiratory disease, reactive airway disease, hepatic or renal disorders.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-10-18 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Ease of successful intubation | Immediately after intubation
  Ease of successful intubation will be measured by the composite score which is a composite of five parameters with a score of 1-5 for each parameter, 1 indicating best possible condition and higher scores indicating worsening of the conditions for intubation . The maximum score was 25. A score of <10 was considered optimal, 10-15

SECONDARY OUTCOMES:
Adverse events. | From intervention for 4hours
  Adverse events (bradycardia, hypotension, laryngeal spasm, lidocaine toxicity). Hypotension (MAP < 20% of baseline readings ). Bradycardia (HR < 50 beats/min
Time till successful intubation. | Immediately after intubation
  Time needed till successful intubation. Direct visualization of the endotracheal tube passing through the vocal cords into the trachea.
Post-operative sore throat. | 24 hours after extubation
  Sore throat will be evaluated at PACU 1, 12 and 24h after extubation, during the post-operative period.
  Grading of Post-operative sore throat (POST) will be done using a four-point scale (0-3) : 0 for no sore throat; 1 for mild sore throat (complains of sore throat only when asked); 2 for moderate sore throat (complains of sore throat even without asking); and 3 for severe sore throat (with change of voice or hoarseness, also may be associated with throat pain).

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author